CLINICAL TRIAL: NCT02994745
Title: A Randomized, Open-label, Single Dose, 3x3 Partial Replicated Crossover Study to Evaluate the Pharmacokinetics and Safety/Tolerability Between a Fixed Dose Combination of Fimasartan 120mg/Atorvastatin 40mg and Co-administration of Fimasartan 120mg and Atorvastatin 40mg in Healthy Male Volunteers.
Brief Title: A Clinical Trial to Evaluate the Pharmacokinetics and Safety/Tolerability of Fimasartan and Atorvastatin in Healthy Male Volunteers.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boryung Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BR-FAVC-CT-102
Record Dates: First submitted 2016-12-01; First posted 2016-12-16 (Estimated); Last update posted 2018-01-18 (Actual); Status verified 2018-01

CONDITIONS: Hypertension, Hyperlipidemia
MeSH Terms: conditions — Hypertension; Hyperlipidemias | interventions — fimasartan; Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A fixed dose combination group (Experimental): A fixed dose combination of Fimasartan/Atorvastatin
  Interventions: Drug: Fimasartan, Atorvastatin
- Co-administration group (Active Comparator): Co-administration of Fimasartan and Atorvastatin
  Interventions: Drug: Fimasartan, Atorvastatin

INTERVENTIONS:
Drug: Fimasartan, Atorvastatin

SUMMARY:
The purpose of this study is to evaluate the Pharmacokinetics and Safety / Tolerability of Fimasartan and Atorvastatin in Healthy Male volunteers.

DETAILED DESCRIPTION:
This is a randomized, open-label, single dose, 3x3 partial replicated crossover study to evaluate the pharmacokinetics and safety/tolerability. Within each period, randomized subjects will be 2 dosing regimens with a fixed dose combination of Fimasartan/Atorvastatin and co-administration of Fimasartan and Atorvastatin.

ELIGIBILITY:
Inclusion Criteria:

* A Healthy male aged 19-50 years
* Body weight is over 55kg and BMI 18 ~ 27(kg/m2).
* A subject provide written informed consent which he voluntarily confirms willingness to participate in a study, having been informed of the full details of the study and comply with the protocol.
* A subject who is eligible according to investigator's assessment

Exclusion Criteria:

* History or presence of clinically significant medical or psychiatric condition or disease.
* History of gastrointestinal disease and resection
* Hypersensitivity to ingredient of investigational product(IP) and other medication, food.
* Genetic Problem such as Galactose intolerance, Lapp lactase deficiency or Glucose-galactose malabsorption.
* A subject who take a drug that inhibit or induce significantly Drug-Metabolizing Enzyme within 1months.
* Positive results for serum examination(HIV, B and C viral test, Syphilis).
* Seated BP is less than 100/65 mmHg or greater than 140/90 mmHg at screening.
* Participation in any other study within 3months.
* History of whole blood donation within 2months and Apheresis 2 weeks.

Ages: 19 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2016-12-23 (Actual); Primary Completion 2017-02-21 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Cmax(Maximum concentration of drug in plasma) of Fimasartan, Atorvastatin | 0~48 hours after medication
AUClast(Area under the plasma drug concentration-time curve over the time interval from 0 to the last quantifiable plasma concentration) of Fimasartan, Atorvastatin | 0~48 hours after medication

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea